CLINICAL TRIAL: NCT05898178
Title: The Effect of Constant 5% Versus Gradient 8%, 5%, 2% Oxygen Concentration on the Development of Sibling Human Embryos in Vitro
Brief Title: Embryo Culture Under Constant 5% vs Gradient 8%, 5%, 2% Oxygen Concentration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Maribor (Other)
Responsible Party: Principal Investigator, Borut Kovačič, Prof. Borut Kovačič, PhD, University Medical Centre Maribor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 0120-405/2021/4; P3-0327 (Other Grant/Funding Number: Slovenian Research Agency)
Record Dates: First submitted 2023-04-26; First posted 2023-06-12 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Embryonic Development; Embryo Morphokinetics; Embryo Morphometry
Keywords: Embryo culture, reduced oxygen, time-lapse, blastocyst

STUDY DESIGN:
Intervention Model Description: 496 sibling oocytes will be randomly allocated for culture either at low oxygen tension (5% O2) (n = 248 oocytes) or a more physiological oxygen gradient (8-5-2% O2) (n = 248 oocytes) for the next 5 days. Immediately after allocation, the oocytes will be inseminated through Intracytoplasmic Sperm Injection (ICSI). The sibling oocytes will always be injected by the same embryologist.
  Under standard (5%) oxygen concentration, which is currently being used in the cultivating incubators, approximately 15% of all embryos manage to reach a morphological optimal blastocyst, in a patient group younger than 35 years (see Inclusion Criteria). According to the hypothesis that cultivating embryos under a more physiological atmosphere (gradient from 8% to 2%) improves the blastulation rate of embryos to 25%, a sample size of 496 Injected oocytes (248 in each arm), will be needed. Whereby a statistical strength of 80% and α = 0.05 is considered (calculated using power analysis).
Who Masked: Investigator
Masking Description: The cohort of oocyte-cumulus complexes will be divided into either the study or control group by simple randomization. All embryologists involved in the study will be blinded during embryo assessment, measurement, and selection for embryo transfer or vitrification. A code system will be used on the Petri dishes to ensure the embryologists are blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 8-5-2% oxygen gradient concentration in the incubator (Experimental): A physiological oxygen gradient concentration in the incubator (8-5-2% O2).
  Interventions: Other: Experimental intervention: 8-5-2% oxygen gradient concentration in the incubator
- Control (no intervention) (No Intervention): Arbitrary cultivation conditions (static 5% 02).

INTERVENTIONS:
Other: Experimental intervention: 8-5-2% oxygen gradient concentration in the incubator — After oocyte retrieval and insemination, half of a given patient's embryos will be randomly allocated in an incubator set at a gradient of oxygen tension (8-5-2%). The embryos will remain in the incubator until their developmental assessments on day 5.
  Arms: 8-5-2% oxygen gradient concentration in the incubator

SUMMARY:
The purpose of this study is to investigate the development of human embryos in vitro under two different oxygen concentrations; a static 5% during all five days of culture or under an oxygen gradient, starting with 8% from day-0 to day-3, continuing with 5% on day-3 and following with 2% of oxygen from the end of day-3 to day-5.

DETAILED DESCRIPTION:
Several studies have shown that embryonic morphological parameters improved when the oxygen concentration in embryo culture was reduced from 20% to 5%. Early mammalian embryos developed faster, had shorter cell cycles, a higher blastocyst formation rate and a better integrity of the inner cell mass (ICM) compared to embryos cultured at 20% oxygen concentration.

Recent studies have shown that the oxygen concentration in the female reproductive tract is not static. In the fallopian tubes of higher mammals it is at around 8%, while in the uterus, at the time of embryo implantation, the oxygen concentration is almost anoxic (2%).

Mimicking such physiological conditions that better reflect the in vivo environment in the human reproductive tract is the goal of assisted reproductive technology (ART).

The aim of this study is to assess whether changing the static 5% oxygen during five days of in vitro embryo culture to the gradient of oxygen, starting with 8% from day-0 to day-3, continuing with 5% on day-3 and following with 2% of oxygen from the end of day-3 to day-5, better reflects conditions found within the human reproductive tract and improves embryo developmental characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Age of women between 18 and 35 years.
* Body mass index (BMI) between 18 and 30 kg/m².
* Only patients with ICSI procedure (male factor of infertility, excluding azoospermia) and blastocyst culture.
* Patients from first and second ICSI cycle attempt.
* Gonadotropin hormone-releasing hormone (GnRH) antagonist cycles.

Exclusion Criteria:

* Presence of endometriosis.
* Previous clinical intervention on ovaries.
* Connected endocrine or metabolic diseases.
* Presence of polycystic ovary syndrome.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 44 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Maribor, Maribor, Slovenia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between January 2022 and January 2023 at the University Medical Centre Maribor. Women under 35 undergoing ICSI for male infertility were included. All patients provided informed consent. A total of 44 participants were enrolled, with a total of 658 cumulus-oocyte complexes (COCs) collected.
Pre-assignment Details: Following oocyte pickup, 625 cumulus-oocyte complexes from 44 ICSI cycles were allocated to two groups by quasi randomisation. After excluding immature (GV/MI) or degenerated oocytes, 521 metaphase II (MII) oocytes remained, with 258 assigned to the control group (5% O₂) and 263 to the intervention group (8-5-2% O₂).
Units Other Than Participants: Injected sibling MII oocytes
Groups:
- 8-5-2% Oxygen Gradient Concentration in the Incubator: The intervention group simulated a dynamic oxygen gradient designed to mimic reported conditions found in vivo, with gas concentrations adjusted according to embryonic developmental stages. From Day 0 to Day 3, the culture environment was set to 6% CO₂, 8% O₂, and 86% N₂. On Day 3, the oxygen concentration was reduced to 5% (6% CO₂, 5% O₂, 89% N₂), and from the end of Day 3 through Day 5, it was further lowered to 2% (6% CO₂, 2% O₂, 92% N₂).
- Control (no Intervention): The control group was maintained under fixed atmospheric conditions with 5% O₂ (6% CO₂, 5% O₂, 89% N₂) throughout the entire culture period, reflecting an arbitrarily used static oxygen culture system.
Period: Overall Study
Arm/Group | 8-5-2% Oxygen Gradient Concentration in the Incubator | Control (no Intervention)
Started | 44; 263 Injected sibling MII oocytes (This was a sibling split-oocyte study, with 44 participants included in both arms, as the same cohort was used-resulting in 44 patients total, not 88.) | 44; 258 Injected sibling MII oocytes (This was a sibling split-oocyte study, with 44 participants included in both arms, as the same cohort was used-resulting in 44 patients total, not 88.)
Completed (As a sibling oocyte study, individual patients were not assigned to different arms; instead, their sibling oocytes were split between the intervention and control groups, allowing direct comparison within the same patient.) | 44; 263 Injected sibling MII oocytes | 44; 258 Injected sibling MII oocytes
Not Completed | 0; 0 Injected sibling MII oocytes | 0; 0 Injected sibling MII oocytes

BASELINE CHARACTERISTICS:
Population: As a sibling oocyte study, individual patients were not assigned to groups; instead, all 44 enrolled female patients had their sibling oocytes allocated between the intervention and control conditions. Thus, a single cohort of patients served as the baseline population.
Groups:
- All Study Participants: As a sibling oocyte study, individual patients were not assigned to groups; instead, all 44 enrolled female patients had their sibling oocytes allocated between the intervention and control conditions. Thus, a single cohort of patients served as the baseline population.
Arm/Group | All Study Participants
Number analyzed (Participants) | 44
Age, Continuous [Median (Standard Deviation); unit: Years] — As a sibling oocyte study, individual patients were not assigned to groups; instead, all 44 enrolled patients had their sibling oocytes allocated between the intervention and control conditions. Thus, a single cohort of patients served as the baseline population.
  Years | 31.4 (2.36)
Sex: Female, Male [Count of Participants; unit: Participants] — As a sibling oocyte study, all 44 enrolled patient couples (each consisting of a female and male partner) participated, but only the female partners' oocytes were allocated between the intervention and control conditions. Therefore, the analysis focuses solely on the female population, with one shared baseline cohort.
  Participants
    Female | 44
    Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Inseminated Oocytes Developed to the Morphologically Optimal Blastocysts on Day 5
Description: The primary outcome measure will be the proportion of oocytes that will develop to the morphologically optimal day-5 blastocysts, scored 4-5AA according to Gardner criteria. According to the scoring system of Gardner, blastocyst morphology parameters such as the degree of blastocoel expansion (1-5), the morphological appearance of the inner cell mass (ICM) (A, B, C) and the cohesiveness of trophectoderm (TE) (A, B, C) will be measured.
Time Frame: Embryos will be annotated on day 5 post insemination (at 8:00 am).
Population: The primary outcome measure is the proportion of inseminated MII oocytes that develop into morphologically optimal day-5 blastocysts, defined as grade 4-5AA according to the Gardner criteria and not the enrolled patient coupled (n=44)
Measure: Number; unit: Oocytes
Units Other Than Participants: Injected metaphase II [MII] oocytes
Arm/Group | 8-5-2% Oxygen Gradient Concentration in the Incubator | Control (no Intervention)
Number analyzed (Participants) | 44 | 44
Number analyzed (Injected metaphase II [MII] oocytes) | 263 | 258
Oocytes | 27 | 38

2. Secondary Outcome: Measured Times From Insemination to Different Embryonic Stages Reached
Description: Using time-lapse software, embryo development videos were reviewed by manually advancing the images frame by frame. Morphokinetic timings were recorded continuously (every 5 minutes) throughout embryo culture, up to 124 hours (Day 5) post-insemination. The following developmental milestones were recorded for each clinically used embryo that reached the blastocyst stage (cryopreserved or transferred):
  tPNa - Appearance of individual pronuclei
  t2 - Time to 2-cell stage
  t3 - Time to 3-cell stage
  t4 - Time to 4-cell stage
  t5 - Time to 5-cell stage
  t6 - Time to 6-cell stage
  t7 - Time to 7-cell stage
  t8 - Time to 8-cell stage
  tSC - First evidence of compaction
  tM - Completion of the compaction process (morula stage)
  tSB - Initiation of blastulation
  tB - Full blastocyst (last frame before zona pellucida starts to thin)
  tEB - Initiation of blastocyst expansion (first frame showing zona thinning)
Time Frame: Morphokinetic timings were recorded continuously (every 5 minutes) throughout embryo culture, up to 124 hours (Day 5) post-insemination.
Population: Embryos included in the analysis were those that progressed to the blastocyst stage and were deemed suitable for clinical use, either through transfer or cryopreservation.
Measure: Median (Inter-Quartile Range); unit: Hours post-insemination (HPI)
Units Other Than Participants: Clinically utilized embryos
Arm/Group | 8-5-2% Oxygen Gradient Concentration in the Incubator | Control (no Intervention)
Number analyzed (Participants) | 44 | 44
Number analyzed (Clinically utilized embryos) | 97 | 122
Hours post-insemination (HPI)
  tPNa | 11.4 [11 to 12.8] | 11.7 [11.1 to 12.6]
  t2 | 25.7 [23.6 to 27.7] | 25.7 [24.9 to 28.5]
  t3 | 36.6 [31.8 to 39.0] | 35.1 [31.7 to 39.2]
  t4 | 38.8 [35.4 to 41.3] | 37.6 [36.0 to 41.0]
  t5 | 49.5 [46.1 to 53.0] | 48.1 [45.0 to 51.3]
  t6 | 53.2 [50.5 to 57.7] | 53.1 [50.3 to 57.7]
  t7 | 61.5 [55.7 to 67.6] | 63.4 [56.8 to 67.8]
  t8 | 69.5 [65.8 to 74.6] | 71.9 [66.4 to 75.1]
  tSC | 86.0 [78.5 to 89.5] | 83.8 [79.0 to 87.5]
  tM | 91.2 [86.8 to 96.5] | 88.3 [84.4 to 92.8]
  tSB | 106.1 [101.4 to 111.1] | 100.8 [96.0 to 106.6]
  tB | 112.4 [108.6 to 117.0] | 106.9 [103.4 to 110.3]
  tEB | 117.0 [115.0 to 122.4] | 111.4 [108.4 to 114.1]

3. Secondary Outcome: Blastocyst and Inner Cell Mass (ICM) Surface Area Measurement on Day 5
Description: Surface measurements of blastocysts and inner cell mass (ICM) will be recorded on time-lapse photos at 116 hours after insemination. The surfaces will be measured in square micrometres using the Primo vision software's measuring tool. An ellipse will be generated around the trophectoderm's outer edge or the inner cell mass. These measurements will exclude the zona pellucida. The measurements will be taken at the focus plane with the largest surface area.
Time Frame: Fix time (116 hours) post insemination
Population: Blastocysts graded Gardner ≥3 were included, as they exhibited sufficient morphological development for accurate measurement of blastocyst and inner cell mass (ICM) surface areas.
Measure: Mean (Standard Deviation); unit: µm²
Units Other Than Participants: Blastocysts graded Gardner ≥ 3
Arm/Group | 8-5-2% Oxygen Gradient Concentration in the Incubator | Control (no Intervention)
Number analyzed (Participants) | 44 | 44
Number analyzed (Blastocysts graded Gardner ≥ 3) | 72 | 110
µm²
  Blastocyst surface area (P, µm²) | 25994 (4657) | 28198 (4139)
  Inner cell mass surface area (ICM, µm²) | 3695 (732.5) | 3628 (831.9)

4. Secondary Outcome: Number of Trophectoderm Cells on Day 5
Description: At 116 hours following insemination, the number of trophectoderm cells will be counted using time-lapse photos. Images will be focused on the trophectoderm's outermost edge to better determine the boundaries of each individual cell.
Time Frame: Fix time (116 hours) post insemination.
Population: Blastocysts graded Gardner ≥3 were included, as these embryos exhibited sufficient morphological development to enable accurate count of trophectoderm (TE) cell number.
Measure: Mean (Standard Deviation); unit: Number of cells
Units Other Than Participants: Blastocysts graded Gardner ≥3
Arm/Group | 8-5-2% Oxygen Gradient Concentration in the Incubator | Control (no Intervention)
Number analyzed (Participants) | 44 | 44
Number analyzed (Blastocysts graded Gardner ≥3) | 72 | 110
Number of cells | 14.4 (2.3) | 15.3 (2.8)

5. Secondary Outcome: Incidence of Atypical Embryo Cleavages
Description: Time-lapse videos for each embryo will be reviewed for atypical cleavage features, such as; pseudofurrows, direct cleavage, reverse cleavage, multinucleation, irregular chaotic division, cell exclusion and blastocyst collapse, using Primo vision software by manually forwarding the images frame by frame. The frequency of abnormal cleavage patterns will be recorded.
Time Frame: Continuously (a picture will be taken every 5 minutes) during 5 days of embryo culture.
Population: The analysis included all embryos that progressed to the blastocyst stage.
Measure: Number; unit: Number of events
Units Other Than Participants: Embryos reaching blastocyst stage
Arm/Group | 8-5-2% Oxygen Gradient Concentration in the Incubator | Control (no Intervention)
Number analyzed (Participants) | 44 | 44
Number analyzed (Embryos reaching blastocyst stage) | 130 | 141
Number of events
  Pseudofurrows | 36 | 49
  Direct cleavage | 25 | 30
  Reverse cleavage | 14 | 9
  Irregular chaotic division | 21 | 15
  Blastomere exclusion | 45 | 34
  Blastocyst collapse | 55 | 67

ADVERSE EVENTS:
Time Frame: No adverse event data were collected from participants. The study focused exclusively on in vitro embryo development. Therefore, no adverse event time frame applies.
Description: Adverse events were not collected, as no participant-level medical events were recorded. The study involved a laboratory-based embryo culture protocol and monitored oocyte/embryo development, not clinical outcomes in patients.
Arm/Group | 8-5-2% Oxygen Gradient Concentration in the Incubator | Control (no Intervention)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-04-24): https://cdn.clinicaltrials.gov/large-docs/78/NCT05898178/Prot_SAP_ICF_000.pdf